CLINICAL TRIAL: NCT05626491
Title: Evaluate the Safety and Efficacy of Repetitive, Transorbital Alternating Current Stimulation (rtACS) for the Treatment of Glaucoma
Brief Title: Electrical Stimulation for the Treatment of Glaucoma
Acronym: rtACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: NYU Langone Health (Other); Otto-von-Guericke University Magdeburg (Other); Wills Eye (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58329
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma; Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active SAVIR Alpha Synch Mobile device (SASm) (Experimental): Patients will receive active treatment with the device every other day over 8 weeks.
  Interventions: Device: Repetitive, Transorbital Alternating Current Stimulation (rtACS)
- Sham SAVIR Alpha Synch Mobile device (SASm) (Sham Comparator): Patients will receive sham treatment (no active stimulation) with the device every other day over 8 weeks.
  Interventions: Device: Sham Repetitive, Transorbital Alternating Current Stimulation (rtACS)

INTERVENTIONS:
Device: Repetitive, Transorbital Alternating Current Stimulation (rtACS) — Patients receive treatment every other day via a headband that delivers electrical stimulation to the retina
  Other Names: Electrical Stimulation
  Arms: Active SAVIR Alpha Synch Mobile device (SASm)
Device: Sham Repetitive, Transorbital Alternating Current Stimulation (rtACS) — Patients receive sham treatment (no active stimulation) every other day via a headband.
  Arms: Sham SAVIR Alpha Synch Mobile device (SASm)

SUMMARY:
The overall aim of this study is to see whether long-term electrical stimulation with a home-stimulation device works well and is safe for the treatment of open-angle glaucoma. Open-Angle Glaucoma is a disease where the nerves in the back of your eye die off faster than expected regardless of your eye pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18.
2. Participant must has the ability to comply with the requirements of the study and complete the schedule of events (SOE).
3. Participant's clinical diagnosis must be consistent with glaucoma characterized by the following features: Mean deviation (MD) worse than -3 on Humphrey Visual Field 24-2 testing. Reliable visual field measures, fixation losses do not exceed 20% and false positives do not exceed 20%.
4. Visual Field Index between 10 and 90%
5. Corrected visual acuity ≥ 1.00 (logMAR), 20/200 (Snellen), 0.10 (decimal)
6. In the opinion of the investigator the participant's eye pressure must be clinically stable.
7. If a participant has two eyes meeting study criteria, the worse eye as determined by mean deviation. If both eyes qualify and have the same MD, the patient may choose which eye they are willing to enter, or else a randomization procedure will assign one eye to the study.
8. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.

Exclusion Criteria:

1. Participant is unable to comply with study procedures or follow-up visits.
2. Participant has a history of ocular herpes zoster.
3. Participant has pathological nystagmus
4. Participant has evidence of visually significant retinopathy including but not limited to Diabetic retinopathy or retinitis pigmentosa.
5. Participant has evidence of corneal opacification or lack of optical clarity.
6. Participant has uveitis or other ocular inflammatory disease.
7. Participant has any electric or electronic implants such as a pacemaker.
8. Participant has acute conjunctivitis.
9. Participant has acute autoimmune disease.
10. Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a drug by ocular (if in the study eye) or systemic administration.
11. Participant is pregnant or lactating.
12. Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments. Including but not limited to all forms of dementia.
13. Unresected brain tumors
14. Implanted intracranial magnetic metals (metallic implants in the head / skull such as clamps, coils, ventriculo-peritoneal shunts, endoprostheses, etc.), which are not MRI-compatible. Note: metallic dental implants and titanium screws or plates are acceptable
15. Patients with any skin damage.
16. Children and comatose patients.
17. Patients with history of epileptic seizure within the last 10 years.
18. Patients with uncontrolled systemic hypertension or uncontrolled diabetes.
19. Self-reported alcohol or illicit drug addictions within the last 12 months.
20. Participant is not able to travel, to comply with the requirements of the study or not willing to complete the schedule of events (SOE) and/or unable to confirm follow-up participation
21. Prior participation in a vision training/stimulation study in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual field assessed by Humphrey Visual Field Index (VFI). | Baseline through 6 months

SECONDARY OUTCOMES:
Change from baseline in visual field assessed by Humphrey Mean Deviation (MD). | Baseline through 6 months
Change from baseline in visual field assessed by Pelli-Robson Contrast Sensitivity. | Baseline through 6 months
  Pelli-Robson is a standard for measuring contrast sensitivity. It is measured on a 0-16 scale. Normal contrast sensitivity is between 12 and 14 with 0 being worst and 16 being best.
Change from baseline in visual acuity as assessed by the Snellen visual acuity test. | Baseline through Month 6
  The Snellen test is a standard eye chart test used to test eyesight.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD PhD, Principal Investigator — Stanford University; Bernhard Sable, PhD, Principal Investigator — Otto-von-Guericke University Magdeburg; Joeseph F Panarelli, MD, Principal Investigator — NYU- Langone; Joel Schuman, MD,FACS, Principal Investigator — Wills Eye
Locations (4):
- United States (3):
  - Byers Eye Institute, Palo Alto, California
  - NYU- Langone, New York, New York
  - Wills Eye Hospital, Philadelphia, Pennsylvania
- Otto-von-Guericke University, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: No